CLINICAL TRIAL: NCT06658912
Title: Planning Grant for Take Off Pounds Sensibly (TOPS) Classes for Breast Cancer Survivors
Brief Title: Planning Grant for TOPS for Breast Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00116571
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Weight Loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOPS Classes (Other)
  Interventions: Other: TOPS Classes

INTERVENTIONS:
Other: TOPS Classes — Attend Dietician-Led Sessions

SUMMARY:
The purpose of this study is to help make a community led weight loss program known as Take Off Pounds Sensibly (TOPS) more relevant for breast cancer survivors.

This study is made up to two parts. The first part includes using focus groups to review current materials that the investigators plan to use in upcoming TOPS classes and provide feedback. Focus groups will be made up of women who are breast cancer survivors.

The second part includes taking the feedback received from these focus groups and use this feedback to tailor TOPS classes for breast cancer survivors.

This ClinicalTrials.gov record is specific to the second part of the study.

DETAILED DESCRIPTION:
The purpose of this study is to help make a community led weight loss program known as Take Off Pounds Sensibly (TOPS) more relevant for breast cancer survivors.

This study is made up to two parts. The first part includes using focus groups to review current materials that the investigators plan to use in upcoming TOPS classes and have the groups provide feedback. Focus groups will be made up of breast cancer survivors that have recruited from local support group chapters. The goal is to recruit approximately 25 people to take part in these focus groups. Meetings of focus groups will be conducted remotely through Zoom and will be recorded. A meeting of the focus group will last anywhere from 60-90 minutes.

The information gathered from these groups will be used to improve the materials which lead to part two of the study.

The second part includes using these materials in TOPS classes that are tailored for breast cancer survivors and determining if the TOPS classes are effective on those who attend the classes. Effectiveness of the class will be determined by the weight loss of the participant and an impact on their heart health.

For the first 6 months, participants will attend dietician-led TOPS sessions conducted virtually through Zoom. Participants' weight will be measured as instructed using a Bluetooth scale that will send their weight measurements back to the team. Participants will also measure their blood pressure through a Bluetooth device provided by the study team.

After 6 months, participants will be asked to join a TOPS chapter in their community. The study team will help them local a chapter that is convenient for them. They must attend these classes for another 6 months. Total time in this portion of the study will be approximately 12 months.

While on study, in addition to measuring their weight and blood pressure via the Bluetooth devices, the study team asks that participants also have their blood collected. Participants will have to go to their local LabCorp facility to have blood drawn at baseline visit, 3 months, 6 months, and 12 months. Participants will also be asked to complete surveys via their email. Surveys will ask about participant's current medications and ask them to score their overall health at that time.

This ClinicalTrials.gov record is specific to the second part of the study.

ELIGIBILITY:
Aim 2 Inclusion Criteria:

* women diagnosed with breast cancer with BMI ≥ 25 kg/m2 after completion of primary therapy (surgery, radiation, adjuvant or neo-adjuvant chemotherapy).

Aim 2 Exclusion Criteria:

* Those whose oncology providers do not agree with their participation in a weight loss program
* History of Type II Diabetes Mellitus
* those participating in another weight loss program
* those taking a weight loss medication
* those without smart phones or internet connections or the ability to attend meetings via Zoom

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of invitations sent through the electronic health record to get 25 individuals consented to the study | 1-2 months
Percentage of TOPS group session attendance | 12 months
  This will be calculated as number of sessions attended divided by total number of sessions offered
Number of participants who stay in the study | 3 months, 6 months, 9 months, 12 months
Number of participants who transition from the initiation phase to the maintenance phase | 12 months
Number of participants who continue to transmit weight and BP data once they transition to the maintenance phase | 9 months, 12 months
Percent of Weight Loss | Up to 12 Months

SECONDARY OUTCOMES:
Cardiovascular Disease (CVD) risk factors as measured by blood pressure | up to 12 months
Cardiovascular Disease (CVD) risk factors as measured by hemoglobin A1c | up to 12 months
Cardiovascular Disease (CVD) risk factors as measured by glucose | up to 12 months
Percentage of participants who get blood drawn | Baseline, 3 months, 6 months,12 months
Quality of Life (QOL) as measured by survey | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nia S Mitchell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No